CLINICAL TRIAL: NCT03023904
Title: Nivolumab in Treating Patients With Stage IV or Recurrent Lung Cancer With High Mutation Loads
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Research cancelled
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Douglas Johnson, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 16117; NCI-2017-00047 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1. Courses repeat every 2 weeks for up to 2 years (104 weeks) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Nivolumab — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well nivolumab works in treating patients with stage IV lung cancer or that has come back after initial treatment who has high mutation loads. Monoclonal antibodies, such as nivolumab, may block tumor growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the objective response rate using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

SECONDARY OBJECTIVES:

I. To assess the progression-free survival (PFS). II. To assess the overall survival (OS). III. To correlate response and mutation load with PD-L1 status (5% and 1% cutoffs).

IV. To assess clinical benefit (responses and stable disease lasting >= 6 months).

V. To assess the response rate in mutation-defined subgroups, including subjects with >= 25 mutations/mutational burden (MB) and >= 30 mutations/MB.

VI. To correlate the type of mutations with response.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 2 weeks for up to 2 years (104 weeks) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 35 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* • Signed written informed consent

  * Subjects must have signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent form in accordance with regulatory and institutional guidelines; this must be obtained before the performance of any protocol related procedures that are not part of normal subject care
  * Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing

    * Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
    * Subjects with histologically confirmed stage IV or recurrent NSCLC (per the 7th International Association for the Study of Lung Cancer classification squamous or nonsquamous histology, with no prior systemic anticancer therapy (including EGFR and ALK inhibitors) given as primary therapy for advanced or metastatic disease
  * Prior adjuvant or neoadjuvant chemotherapy is permitted as long as the last administration is at least 2 months prior to enrollment
  * Prior definitive chemoradiation for locally advanced disease is also permitted as long as the last administration of chemotherapy or radiotherapy (whichever was given last) occurred at least 2 months prior to enrollment

    * Mutation load determined by FoundationOne of >= 20 mutations/MB tested on archival tumor sample; the mutation load metric will be displayed on the FoundationOne report for all participating sites as "tumor mutation burden (TMB) - high" or may be obtained from Foundation Medicine from older reports using the Insights Portal, which will be available to all participating sites, or by emailing Foundation Medicine
    * Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1 criteria
  * Target lesions may be located in a previously irradiated field if there is documented (radiographic) disease progression in that site after the completion of radiation therapy

    * Prior palliative radiotherapy to non-central nervous system (CNS) lesions must have been completed at least 2 weeks prior to enrollment; subjects with symptomatic tumor lesions at baseline that may require palliative radiotherapy within 4 weeks of enrollment are strongly encouraged to receive palliative radiotherapy prior to enrollment
    * White blood cell (WBC) > 2000/uL
    * Neutrophils > 1500/uL
    * Platelets > 100 x 10^9/uL
    * Hemoglobin > 9.0 g/dL
    * Serum creatinine =< 2 x upper limit normal (ULN) or creatinine clearance (CrCl) >= 30 mL/min using the Cockcroft-Gault formula
    * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN (unless liver metastases, who can have AST/ALT =< 5 x ULN)
    * Total bilirubin =< 3 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
    * Women must not be breastfeeding
    * Women of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to the start of nivolumab
  * "Women of childbearing potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal
  * Menopause is defined as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; if menopausal status is considered for the purpose of evaluating childbearing potential, women under the age of 62 must have a documented serum follicle stimulating hormone (FSH) level > 40 mIU/mL, in order to be considered postmenopausal and not of childbearing potential

    • Women of child bearing potential (WOCBP) and men able to father children who are sexually active with WOCBP must agree to use acceptable contraception
  * Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) and azoospermic men do not require contraception
  * Women of childbearing potential receiving nivolumab will be instructed to use and must be willing to use appropriate method(s) of contraception for a period of 23 weeks after the last dose of investigational product
  * Men receiving nivolumab who are sexually active with WOCBP will be instructed to use and must be willing to use acceptable contraception for a period of 31 weeks after the last dose of investigational product

Exclusion Criteria:

* Subjects with known EGFR mutations which are sensitive to available targeted inhibitor therapy (including, but not limited to, deletions in exon 19 and exon 21 [L858R] substitution mutations) are excluded; all subjects with non-squamous histology must have been tested for EGFR mutation status; use of a Food and Drug Administration (FDA)-approved test is strongly encouraged
* Subjects with known ALK translocations which are sensitive to available targeted inhibitor therapy are excluded; if tested, use of an FDA-approved test is strongly encouraged; subjects with unknown or indeterminate ALK status may be enrolled
* Active brain metastases or leptomeningeal metastases (carcinomatous meningitis); subjects with brain metastases are eligible if these have been treated and there is no evidence of progression for at least 2 weeks after treatment is complete and corticosteroid dose is stable (and equivalent dose of < 10 mg prednisone) for at least 2 weeks
* Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before enrollment
* Subjects with an active, known or suspected autoimmune disease; subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first study treatment with nivolumab; inhaled or topical steroids, and adrenal replacement steroid > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Patients with concurrent severe and/or uncontrolled concurrent medical conditions that could compromise participation in the study (e.g., uncontrolled hypertension and/or diabetes mellitus, clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection)
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration
* Subjects with previous or active malignancies (except non-melanoma skin cancers, and in situ cancers such as the following: bladder, gastric, colon, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to enrollment and no additional therapy is required or anticipated to be required during the study period
* History of allergy to study drug components or of severe hypersensitivity reaction to any monoclonal antibody
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate defined as the number of subjects with a best overall response of complete response or partial response divided by the number of subjects that receive nivolumab as assessed by RECIST 1.1 | Up to 6 months

SECONDARY OUTCOMES:
Overall survival | From date of enrollment to date of death due to any cause, assessed up to 2 years
Progression Free Survival as determined by RECIST 1.1 | From date of enrollment until first date of documented progression or death due to any cause, assessed up to 2 years
Mutation load as determined by FoundationOne testing | Up to 2 years
Incidence of adverse events (AEs) graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Up to 100 days after the last dose of study drug
PD-L1 expression as determined by immunohistochemistry | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Johnson, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center

IPD SHARING:
Plan to Share IPD: Undecided